CLINICAL TRIAL: NCT00575354
Title: Anesthesia With Sevoflurane and Isoflurane for Excision Surgeries in Benign Breast Tumors
Brief Title: Comparison of Sevoflurane and Isoflurane Anesthesia for Benign Breast Tumor Excision
Acronym: CSIABTEC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMU-2579-6FW; #NMU072036
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Breast Neoplasms
Keywords: Sevoflurane; Isoflurane; Breast tumor; Anesthesia
MeSH Terms: conditions — Breast Neoplasms | interventions — Sevoflurane; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Sevoflurane: induction 3-6%, maintenance 2-3%
  Interventions: Drug: Sevoflurane
- 2 (Active Comparator): Isoflurane: induction 3-6%, maintenance 2-3%
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Sevoflurane — 3-6% sevoflurane inhaled for anesthesia induction, and 2-3% sevoflurane was used to maintain the anesthesia till the end of the operation.
  Other Names: Sevofrane
  Arms: 1
Drug: Isoflurane — 3-6% isoflurane inhaled for anesthesia induction, and 2-3% isoflurane was used to maintain the anesthesia till the end of the operation.
  Arms: 2

SUMMARY:
Generally, benign breast tumors are excised under the local anesthesia. But such action was so invasive that every patient would experience the physiological and psychological stimuli unavoidably. Sevoflurane was advised as a better inhalational anesthesic for its "easy come,easy go" property during short-lasting operations than isoflurane. We purposed that sevoflurane would be a superior anesthesic for benign breast tumor excision than isoflurane with relative less alteration in hemodynamics, less postoperative side effects and easily-control the depth of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Chinese
* Diagnosed benign breast tumor patients
* 18-64 yrs

Exclusion Criteria:

* Allergic to any interventional drugs
* Organic dysfunction
* Long-lasting PACU staying

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Time of induction, maintenance and resuscitation | 0h to the end of the operation

SECONDARY OUTCOMES:
Intraoperative hemodynamics; Postoperative side effects; | 0h to 24h after the end of the operation

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Care Hospital, Nanjing, Jiangsu, China